CLINICAL TRIAL: NCT03896581
Title: A Multicenter, Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Bimekizumab in the Treatment of Subjects With Active Psoriatic Arthritis
Brief Title: A Study to Evaluate the Efficacy and Safety of Bimekizumab in the Treatment of Subjects With Active Psoriatic Arthritis
Acronym: BE COMPLETE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PA0011; 2017-002804-29 (EudraCT Number)
Record Dates: First submitted 2019-03-21; First posted 2019-04-01 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; PsA; Bimekizumab
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimekizumab dosage regimen (Experimental): Subjects randomized to this arm will receive assigned bimekizumab dosage regimen.
  Interventions: Drug: Bimekizumab
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive bimekizumab at pre-specified time-points.
  Other Names: BKZ; UCB4940
  Arms: Bimekizumab dosage regimen
Other: Placebo — Subjects will receive placebo at pre-specified time-points.
  Other Names: PBO
  Arms: Placebo

SUMMARY:
This is a study to demonstrate the clinical efficacy, safety and tolerability of bimekizumab administered subcutaneously (sc) compared with placebo in the treatment of tumor necrosis factor alpha-inadequate responders (TNFα-IR) subjects with active Psoriatic Arthritis (PsA).

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female at least 18 years of age
* Female subjects must be postmenopausal, permanently sterilized or willing to use a highly effective method of contraception
* Documented diagnosis of adult-onset Psoriatic Arthritis (PsA) meeting the Classification Criteria for Psoriatic Arthritis (CASPAR) for at least 6 months prior to Screening with active PsA and must have at Baseline tender joint count (TJC) >=3 out of 68 and swollen joint count (SJC) >=3 out of 66
* Subject must be negative for rheumatoid factor and anti-cyclic citrullinated peptide (CCP) antibodies
* Subject must have at least 1 active psoriatic lesion(s) and/or a documented history of psoriasis (PSO)
* Subject has a history of inadequate response (lack of efficacy after at least 3 months of therapy at an approved dose) or intolerance to treatment with 1 or 2 tumor necrosis factor alpha (TNF(α)) inhibitors for either PsA or PSO
* Subjects currently taking NSAIDs, cyclooxygenase 2 (COX-2) inhibitors, analgesics (including mild opioids), corticosteroids, methotrexate (MTX), leflunomide (LEF), sulfasalazine (SSZ), hydroxychloroquine (HCQ) AND/OR apremilast can be allowed if they fulfill specific requirements prior to study entry

Exclusion Criteria:

* Female subjects who are breastfeeding, pregnant, or plan to become pregnant during the study
* Subjects with current or prior exposure to any biologics except tumor necrosis factor (TNF) inhibitors for the treatment of PsA or PSO
* Subject has an active infection or a history of recent serious infections
* Subject has known tuberculosis (TB) infection, is at high risk of acquiring TB infection, or has current or history of nontuberculous mycobacterium (NTMB) infection
* Subject has a diagnosis of inflammatory conditions other than PSO or PsA. Subjects with a diagnosis of Crohn's disease, ulcerative colitis, or other inflammatory bowel disease (IBD) are allowed as long as they have no active symptomatic disease at Screening or Baseline
* Subject had acute anterior uveitis within 6 weeks of Baseline
* Subject has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, or in situ cervical cancer
* Subject has a form of PSO other than chronic plaque-type (eg, pustular, erythrodermic and guttate PSO, or drug-induced PSO)
* Presence of active suicidal ideation, or moderately severe major depression or severe major depression
* Subject has a history of chronic alcohol or drug abuse within 6 months prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (92):
- United States (33):
  - Pa0011 50017, Phoenix, Arizona
  - Pa0011 50035, San Diego, California
  - Pa0011 50004, Tustin, California
  - Pa0011 50033, Palm Harbor, Florida
  - Pa0011 50037, Tampa, Florida
  - Pa0011 50039, Atlanta, Georgia
  - Pa0011 50024, Boise, Idaho
  - Pa0011 50028, Lexington, Kentucky
  - Pa0011 50023, Baton Rouge, Louisiana
  - Pa0011 50015, Hagerstown, Maryland
  - Pa0011 50026, Wheaton, Maryland
  - Pa0011 50047, Boston, Massachusetts
  - Pa0011 50019, Lansing, Michigan
  - Pa0011 50016, St Louis, Missouri
  - Pa0011 50005, Freehold, New Jersey
  - Pa0011 50029, Albuquerque, New Mexico
  - Pa0011 50010, Brooklyn, New York
  - Pa0011 50011, New York, New York
  - Pa0011 50034, Rochester, New York
  - Pa0011 50125, Charlotte, North Carolina
  - Pa0011 50031, Salisbury, North Carolina
  - Pa0011 50040, Vandalia, Ohio
  - Pa0011 50020, Duncansville, Pennsylvania
  - Pa0011 50064, Philadelphia, Pennsylvania
  - Pa0011 50006, Wyomissing, Pennsylvania
  - Pa0011 50008, Johnston, Rhode Island
  - Pa0011 50021, Summerville, South Carolina
  - Pa0011 50001, Jackson, Tennessee
  - Pa0011 50012, Memphis, Tennessee
  - Pa0011 50002, Austin, Texas
  - Pa0011 50036, Mesquite, Texas
  - Pa0011 50009, Waco, Texas
  - Pa0011 50050, Beckley, West Virginia
- Australia (3):
  - Pa0011 30005, Camberwell
  - Pa0011 30007, Victoria Park
  - Pa0011 30006, Woodville South
- Canada (3):
  - Pa0011 50042, Rimouski
  - Pa0011 50043, Sydney
  - Pa0011 50044, Trois-Rivières
- Czechia (4):
  - Pa0011 40009, Pardubice
  - Pa0011 40063, Prague
  - Pa0011 40066, Prague
  - Pa0011 40012, Zlín
- Germany (7):
  - Pa0011 40076, Cottbus
  - Pa0011 40023, Erlangen
  - Pa0011 40117, Frankfurt
  - Pa0011 40029, Hamburg
  - Pa0011 40071, Hamburg
  - Pa0011 40078, Leipzig
  - Pa0011 40026, Ratingen
- Hungary (2):
  - Pa0011 40083, Budapest
  - Pa0011 40079, Szentes
- Italy (3):
  - Pa0011 40084, Catania
  - Pa0011 40087, Milan
  - Pa0011 40086, Reggio Emilia
- Japan (11):
  - Pa0011 20030, Chūōku
  - Pa0011 20043, Itabashi-ku
  - Pa0011 20036, Kawachi-Nagano
  - Pa0011 20045, Kita-gun
  - Pa0011 20049, Kitakyushu
  - Pa0011 20044, Minatoku
  - Pa0011 20041, Osaka
  - Pa0011 20046, Osaka
  - Pa0011 20031, Sapporo
  - Pa0011 20042, Sasebo
  - Pa0011 20032, Suita
- Poland (12):
  - Pa0011 40119, Bydgoszcz
  - Pa0011 40038, Elblag
  - Pa0011 40037, Lublin
  - Pa0011 40091, Nowa Sól
  - Pa0011 40044, Poznan
  - Pa0011 40090, Poznan
  - Pa0011 40118, Torun
  - Pa0011 40041, Warsaw
  - Pa0011 40097, Warsaw
  - Pa0011 40098, Warsaw
  - Pa0011 40039, Wroclaw
  - Pa0011 40043, Wroclaw
- Russia (11):
  - Pa0011 20005, Korolyov
  - Pa0011 20010, Moscow
  - Pa0011 20013, Petrozavodsk
  - Pa0011 20001, Saint Petersburg
  - Pa0011 20004, Saint Petersburg
  - Pa0011 20009, Saint Petersburg
  - Pa0011 20007, Saratov
  - Pa0011 20014, Ulyanovsk
  - Pa0011 20006, Vladimir
  - Pa0011 20008, Yaroslavl
  - Pa0011 20015, Yaroslavl
- United Kingdom (3):
  - Pa0011 40111, Bradford
  - Pa0011 40109, Oxford
  - Pa0011 40116, Stamford

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Secukinumab in Patients with Psoriatic Arthritis at 52 Weeks Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Jun;11(3):817-828. doi: 10.1007/s40744-024-00652-7. Epub 2024 Mar 6. PMID 38446397
- [Result] Warren RB, McInnes IB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, Mease PJ. Comparative Effectiveness of Bimekizumab and Guselkumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Jun;11(3):829-839. doi: 10.1007/s40744-024-00659-0. Epub 2024 Mar 15. PMID 38488975
- [Result] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Risankizumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Oct;11(5):1403-1412. doi: 10.1007/s40744-024-00706-w. Epub 2024 Aug 9. PMID 39120849
- [Result] Kristensen LE, Tillett W, Nash P, Coates LC, Mease PJ, Ogdie A, Gisondi P, Ink B, Prickett AR, Bajracharya R, Taieb V, Lyris N, Lambert J, Walsh JA. Association of achieving clinical disease control criteria and patient-reported outcomes in bimekizumab-treated patients with active psoriatic arthritis: results from two phase III studies. Ther Adv Musculoskelet Dis. 2024 Nov 11;16:1759720X241288071. doi: 10.1177/1759720X241288071. eCollection 2024. PMID 39534481
- [Result] Mease PJ, Merola JF, Tanaka Y, Gossec L, McInnes IB, Ritchlin CT, Landewe RBM, Asahina A, Ink B, Heinrichs A, Bajracharya R, Shende V, Coarse J, Coates LC. Summary of Research: Safety and Efficacy of Bimekizumab in Patients with Psoriatic Arthritis: 2-Year Results from Two Phase 3 Studies. Rheumatol Ther. 2025 Aug;12(4):609-612. doi: 10.1007/s40744-025-00764-8. Epub 2025 May 10. PMID 40347389
- [Result] Thaci D, Asahina A, Boehncke WH, Gottlieb AB, Lebwohl M, Warren RB, Edens H, Ink B, Bajracharya R, Coarse J, Merola JF. Bimekizumab Efficacy and Safety in Patients with Psoriatic Arthritis with Substantial Skin and Nail Psoriasis to 1 Year. Dermatol Ther (Heidelb). 2025 Dec 12. doi: 10.1007/s13555-025-01599-5. Online ahead of print. PMID 41381988
- [Derived] Mease PJ, Gensler LS, Orbai AM, Warren RB, Bajracharya R, Ink B, Marten A, Massow U, Shende V, Manente M, Peterson L, White K, Landewe R, Poddubnyy D. Long-term safety of bimekizumab in adult patients with axial spondyloarthritis or psoriatic arthritis: pooled results from integrated phase IIb/III clinical studies. RMD Open. 2025 Apr 6;11(2):e005026. doi: 10.1136/rmdopen-2024-005026. PMID 40194794
- [Derived] Gladman DD, Mease PJ, Gossec L, Husni ME, Gottlieb AB, Ink B, Bajracharya R, Coarse J, Lyris N, Lambert J, Tillett W. Effect of Bimekizumab on Patient-Reported Outcomes and Work Productivity in Patients With Psoriatic Arthritis: 1-Year Results From 2 Phase III Studies. J Rheumatol. 2025 May 1;52(5):466-478. doi: 10.3899/jrheum.2024-0923. PMID 39892885
- [Derived] Husni ME, Mease PJ, Merola JF, Tillett W, Goldammer N, Ink B, Coarse J, Lambert J, Taieb V, Gladman DD. Bimekizumab provided rapid improvements in patient-reported symptoms and health-related quality of life in patients with active psoriatic arthritis: pooled 16-week results from two phase 3 studies. RMD Open. 2024 Sep 23;10(3):e004464. doi: 10.1136/rmdopen-2024-004464. PMID 39313302
- [Derived] Mease PJ, Merola JF, Tanaka Y, Gossec L, McInnes IB, Ritchlin CT, Landewe RBM, Asahina A, Ink B, Heinrichs A, Bajracharya R, Shende V, Coarse J, Coates LC. Safety and Efficacy of Bimekizumab in Patients with Psoriatic Arthritis: 2-Year Results from Two Phase 3 Studies. Rheumatol Ther. 2024 Oct;11(5):1363-1382. doi: 10.1007/s40744-024-00708-8. Epub 2024 Aug 31. PMID 39215949
- [Derived] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Ustekinumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Oct;11(5):1413-1423. doi: 10.1007/s40744-024-00705-x. Epub 2024 Aug 9. PMID 39120848
- [Derived] Gossec L, Orbai AM, de Wit M, Coates LC, Ogdie A, Ink B, Coarse J, Lambert J, Taieb V, Gladman DD. Effect of bimekizumab on patient-reported disease impact in patients with psoriatic arthritis: 1-year results from two phase 3 studies. Rheumatology (Oxford). 2024 Sep 1;63(9):2399-2410. doi: 10.1093/rheumatology/keae277. PMID 38754125
- [Derived] Maloney A, Dua P, Ahmed GF. Comparative Effectiveness of Bimekizumab in Psoriatic Arthritis: A Model-Based Meta-Analysis of American College of Rheumatology Response Criteria. Clin Pharmacol Ther. 2024 May;115(5):1007-1014. doi: 10.1002/cpt.3135. Epub 2024 Jan 12. PMID 38073049
- [Derived] Merola JF, Landewe R, McInnes IB, Mease PJ, Ritchlin CT, Tanaka Y, Asahina A, Behrens F, Gladman DD, Gossec L, Gottlieb AB, Thaci D, Warren RB, Ink B, Assudani D, Bajracharya R, Shende V, Coarse J, Coates LC. Bimekizumab in patients with active psoriatic arthritis and previous inadequate response or intolerance to tumour necrosis factor-alpha inhibitors: a randomised, double-blind, placebo-controlled, phase 3 trial (BE COMPLETE). Lancet. 2023 Jan 7;401(10370):38-48. doi: 10.1016/S0140-6736(22)02303-0. Epub 2022 Dec 6. PMID 36495881
- See also: Product Information — https://www.ema.europa.eu/en/documents/product-information/bimzelx-epar-product-information_en.pdf
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in March 2019 and concluded in February 2022.
Pre-assignment Details: Participant Flow refers to the Randomized Set.
Groups:
- Placebo: Participants received placebo as a subcutaneous (sc) injection every 4 weeks (Q4W) for up to 16 weeks.
- Bimekizumab 160mg: Participants received bimekizumab (BKZ) 160 milligrams (mg) as a sc injection Q4W for up to 16 weeks.
Period: Overall Study
Arm/Group | Placebo | Bimekizumab 160mg
Started | 133 | 267
Completed | 125 | 263
Not Completed | 8 | 4
Not completed — Other (Covid-19 Pandemic Circumstances) | 1 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 2 | 1
Not completed — Adverse event, non-fatal | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to Randomized Set which consisted of all enrolled participants who had been randomized.
Groups:
- Placebo: Participants received placebo as a sc injection Q4W for up to 16 weeks.
- Bimekizumab 160mg: Participants received bimekizumab 160 mg as a sc injection Q4W for up to 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Bimekizumab 160mg | Total
Number analyzed (Participants) | 133 | 267 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 111 | 226 | 337
  >=65 years | 22 | 41 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.30 (12.876) | 50.13 (12.382) | 50.52 (12.545)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 137 | 210
  Male | 60 | 130 | 190
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 9 | 13
  White | 128 | 256 | 384
  Other/Mixed | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 130 | 266 | 396

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology 50 (ACR50) Response
Description: The ACR50 response rate was based on a 50% or greater improvement of arthritis relative to Baseline. Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR50 response criteria: 1.≥ 50% improvement in 68-tender joint count; 2.≥ 50% improvement in 66-swollen joint count; and 3.≥ 50% improvement in at least 3 of the 5 following parameters: Physician global assessment of disease activity [100 mm visual analog scale (VAS) (0=no symptoms;100=severe symptoms)], Patient global assessment of disease activity [100 mm VAS (0=no limitation of normal activities;100=very poor], Patient assessment of pain [100 mm VAS (0=no pain;100=most severe pain)], Health Assessment Questionnaire - Disability Index (HAQ-DI) assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), its score (0-3) computed from item scores, lower scores indicated less disability and high-sensitivity C-reactive protein (hsCRP).
Time Frame: From Baseline to Week 16
Population: Randomized Set consisted of all enrolled participants who had been randomized. Participants who had missing ACR50 data at Week 16 or who discontinued study treatment before Week 16 regardless of whether they had data or not are considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 133 | 267
percentage of participants | 6.8 | 43.4
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 160mg; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.139, 95% CI 2-sided [5.402 to 22.969]

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Total Score at Week 16
Description: The HAQ-DI contains 20 items that measured the degree of difficulty experienced in the following 8 categories of the daily living activities: dressing and grooming (2 items), arising (2 items), eating (3 items), walking (2 items), hygiene (3 items), reach (2 items), grip (3 items), and common daily activities (3 items). Each question was scored 0-3 (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do). The overall HAQ-DI total score was calculated by dividing the sum of the highest category scores (0 to 24) by the number of categories with at least 1 question answered. The HAQ-DI score ranges from 0 (no difficulty) to 3 (maximum difficulty). A lower HAQ-DI score indicated an improvement in function. Change from baseline was computed as the value at Week 16 minus the baseline value. A negative value in change from baseline indicated an improvement.
Time Frame: Baseline and Week 16
Population: Randomized Set consisted of all enrolled participants who had been randomized. Missing data and non-missing data preceded by a study treatment discontinuation were imputed using multiple imputation.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 133 | 267
score on a scale | -0.0701 (0.0432) | -0.3751 (0.0286)
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 160mg; Test type: Superiority; p < 0.001, ANCOVA; Least square (LS) mean difference = -0.326, 95% CI 2-sided [-0.420 to -0.233]

3. Secondary Outcome: Psoriasis Area Severity Index 90 Response (PASI90) at Week 4 in the Subgroup of Participants With Psoriasis (PSO) Involving at Least 3% Body Surface Area (BSA) at Baseline
Description: The PASI90 response assessments are based on at least 90% improvement in PASI score from Baseline. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of respective section, and weighted by the percentage of the person's affected skin for respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: From Baseline to Week 4
Population: Subset of study participants in Randomized Set with psoriasis involving at least 3% BSA at Baseline. Participants who had missing PASI90 data at Week 4 or who discontinued study treatment before or at Week 4 regardless whether they had data or not are considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 88 | 176
percentage of participants | 0 | 26.7

4. Secondary Outcome: Psoriasis Area Severity Index 90 (PASI90) Response at Week 16 in the Subgroup of Participants With Psoriasis (PSO) Involving at Least 3% Body Surface Area at Baseline
Description: as for outcome 3
Time Frame: From Baseline to Week 16
Population: Subset of study participants in Randomized Set with psoriasis involving at least 3% BSA at Baseline. Participants who had missing PASI90 data at Week 16 or who discontinued study treatment before or at Week 16 regardless whether they had data or not are considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 88 | 176
percentage of participants | 6.8 | 68.8
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 160mg; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 30.237, 95% CI 2-sided [12.365 to 73.940]

5. Secondary Outcome: Change From Baseline in the Short Form 36-item Health Survey (SF-36) Physical Component Summary (PCS) Score at Week 16
Description: The SF-36 (version 2, standard recall) is a 36-item generic HRQoL instrument that uses a recall period of 4 weeks. The questionnaire has 36 questions composing the scale that represent 8 domains: 1) physical functioning, 2) role physical, 3) bodily pain, 4) general health, 5) vitality, 6) social functioning, 7) role emotional, and 8) mental health. The scores for the 8 domains were combined into two summary scores: the physical component summary (PCS) score and the mental component summary (MCS) score. Domains 1 to 4 primarily contribute to the PCS score of the SF-36. Domains 5-8 primarily contribute to the MCS score of the SF-36. Each of the 8 domain scores and the component summary score range from 0=worst to 100=best. Higher scores represent better health status. A positive change in value indicated improvement from baseline.
Time Frame: Baseline and Week 16
Population: Randomized Set consisted of all enrolled participants who had been randomized.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 133 | 267
score on a scale | 1.413 (0.714) | 7.258 (0.531)
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 160mg; Test type: Superiority; p < 0.001, ANCOVA; LS mean difference = 6.037, 95% CI 2-sided [4.386 to 7.688]

6. Secondary Outcome: Minimal Disease Activity (MDA) at Week 16
Description: MDA is a measure to indicate disease remission, and is based on a composite score of 7 domains. A participant is considered as having achieved the MDA if the participant fulfills at least 5 of the following 7 criteria: Tender joint count (0-68 joints) <=1; Swollen joint count (0-66 joints) <=1; PASI <=1 for participants with psoriasis covering BSA <=3% [PASI evaluates the severity and extent of psoriasis. In PASI, body is divided into four parts, head and neck, upper limb, trunk and lower limbs. Each area is assessed for erythema, induration and scaling, each rated on a scale of 0 to 4. The total score ranges from 0 (no disease) to 72 (maximal disease)]; Patient's Assessment of Arthritis Pain <=15 [using VAS on a scale of 0 (no pain) to 100 (serious pain)]; Patient's Global Assessment of Disease Activity <=20 [using VAS on a scale of 0 (very well) to 100 (very poor)]; HAQ-DI score <=0.5; Leeds Enthesitis Index score <=1 for participants with enthesitis at baseline.
Time Frame: Week 16
Population: Randomized Set consisted of all enrolled participants who had been randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 133 | 267
percentage of participants | 6.0 | 44.2
Statistical Analysis 1: Comparison: Placebo vs Bimekizumab 160mg; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 13.089, 95% CI 2-sided [6.119 to 27.999]

7. Secondary Outcome: Percentage of Participants With American College of Rheumatology 20 (ACR20) Response
Description: The ACR20 response rate was based on a 20% or greater improvement of arthritis relative to Baseline. Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria: 1.≥ 20% improvement in 68-tender joint count; 2.≥ 20% improvement in 66-swollen joint count; and 3.≥ 20% improvement in at least 3 of the 5 following parameters: Physician global assessment of disease activity [100 mm VAS (0=no symptoms;100=severe symptoms)], Patient global assessment of disease activity [100 mm VAS (0=no limitation of normal activities;100=very poor], Patient assessment of pain [100 mm VAS (0=no pain;100=most severe pain)], HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), its score (0-3) computed from item scores, lower scores indicated less disability, hsCRP.
Time Frame: From Baseline to Week 16
Population: Randomized Set consisted of all enrolled participants who had been randomized. Participants who had missing ACR20 data at Week 16 or who discontinued study treatment before Week 16 regardless of whether they had data or not are considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 133 | 267
percentage of participants | 15.8 | 67.0

8. Secondary Outcome: Percentage of Participants With American College of Rheumatology 70 (ACR70) Response
Description: The ACR70 response rate was based on a 70% or greater improvement of arthritis relative to Baseline. Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria: 1.≥ 70% improvement in 68-tender joint count; 2.≥ 70% improvement in 66-swollen joint count; and 3.≥ 70% improvement in at least 3 of the 5 following parameters: Physician global assessment of disease activity [100 mm VAS (0=no symptoms;100=severe symptoms)], Patient global assessment of disease activity [100 mm VAS (0=no limitation of normal activities;100=very poor], Patient assessment of pain [100 mm VAS (0=no pain;100=most severe pain)], HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), its score (0-3) computed from item scores, lower scores indicated less disability, hsCRP.
Time Frame: From Baseline to Week 16
Population: Randomized Set consisted of all enrolled participants who had been randomized. Participants who had missing ACR70 data at Week 16 or who discontinued study treatment before Week 16 regardless of whether they had data or not are considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 133 | 267
percentage of participants | 0.8 | 26.6

9. Secondary Outcome: Investigator Global Assessment (IGA) Response Defined as Score of 0 (Clear) or 1 (Almost Clear) and at Least a 2-grade Reduction From Baseline at Week 4 in the Subset of Participants With Psoriatic Skin Lesions at Baseline
Description: IGA measured the overall severity of PSO using the following 5-point scale and score was rated as 0=clear (No signs of PSO; post-inflammatory hyperpigmentation may be present), 1=almost clear (No thickening; normal to pink coloration; no to minimal focal scaling), 2=mild (Just detectable to mild thickening; pink to light red coloration; predominately fine scaling), 3=moderate (Clearly distinguishable to moderate thickening; dull to bright red, moderate scaling), and 4=severe (Severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions). The IGA response is defined as score of 0 (clear) or 1 (almost clear) with at least a 2-category improvement relative to Baseline.
Time Frame: Baseline and Week 4
Population: Subset of study participants in Randomized Set with psoriatic skin lesions at Baseline. Participants who had missing data at the Week 4 or who discontinued study treatment before or at the Week 4 regardless whether they had data or not are considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 82 | 163
percentage of participants | 1.2 | 30.7

10. Secondary Outcome: Investigator Global Assessment (IGA) Response Defined as Score of 0 (Clear) or 1 (Almost Clear) and at Least a 2-grade Reduction From Baseline at Week 16 in the Subset of Participants With Psoriatic Skin Lesions at Baseline
Description: as for outcome 9
Time Frame: Baseline and Week 16
Population: Subset of study participants in Randomized Set with psoriatic skin lesions at Baseline. Participants who had missing data at the Week 16 or who discontinued study treatment before or at the Week 16 regardless whether they had data or not are considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 82 | 163
percentage of participants | 3.7 | 60.7

11. Secondary Outcome: Change From Baseline in the Patient's Assessment of Arthritis Pain (PtAAP) at Week 16
Description: The PtAAP Visual Analog Scale (VAS) is part of the American College of Rheumatology core set of measures in arthritis. Participants assessed their arthritis pain using a VAS on a scale of 0 (very well) to 100 (very poor). A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: Randomized Set consisted of all enrolled participants who had been randomized.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 133 | 267
score on a scale | -4.5 (2.1) | -27.7 (1.7)

12. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Impact of Disease-12 (PsAID-12) Total Score at Week 16
Description: The PsAID-12 is a patient-reported outcome measure for assessing the impact of Psoriatic Arthritis (PsA) in 12 physical and psychological domains, including pain, fatigue, skin problems, work and/or leisure activities, functional capacity, discomfort, sleep disturbance, coping, anxiety/fear/uncertainty, embarrassment and/or shame, social participation, and depression. Each domain is assessed with a single question using a 0 to 10 numerical rating scale. Each domain score was multiplied by a weighting factor and the results were then summed to provide the total score. The total score ranged from 0 to 10, with higher scores indicating a worse status. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: Randomized Set consisted of all enrolled participants who had been randomized.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 133 | 267
score on a scale | -0.32 (0.16) | -2.24 (0.13)

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) During the Study
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAEs were defined as any AEs with an onset date on or after the date of first IMP administration and up to 20 weeks after the last (most recent) dose of IMP.
Time Frame: From Baseline until Safety Follow-Up (up to 37 weeks)
Population: The Safety Set consisted of all participants who received at least 1 dose of the IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 132 | 267
Participants | 44 | 108

14. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs) During the Study
Description: A serious adverse event (SAE) is any untoward medical occurrence that at any dose: Results in death, Is life-threatening, Requires in patient hospitalization or prolongation of existing hospitalization; Is a congenital anomaly or birth defect; Is an infection that requires treatment parenteral antibiotics, Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above. TEAEs were defined as any AEs with an onset date on or after the date of first IMP administration and up to 20 weeks after the last (most recent) dose of IMP.
Time Frame: From Baseline until Safety Follow-Up (up to 37 weeks)
Population: The Safety Set consisted of all participants who received at least 1 dose of the IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 132 | 267
Participants | 0 | 5

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Withdrawal From Investigational Medicinal Product (IMP) During the Study
Description: as for outcome 13
Time Frame: From Baseline until Safety Follow-Up (up to 37 weeks)
Population: The Safety Set consisted of all participants who received at least 1 dose of the IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bimekizumab 160mg
Number analyzed (Participants) | 132 | 267
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: From Baseline until Safety Follow-Up (up to 37 weeks)
Description: Treatment-emergent adverse events (TEAEs) were defined as any AEs with an onset date on or after the date of first IMP administration and up to 20 weeks after the last (most recent) dose of IMP. TEAEs were analyzed for Safety Set.
Arm/Group | Placebo | Bimekizumab 160mg
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/267
Serious Adverse Events (participants affected / at risk) | 0/132 | 5/267
Other Adverse Events (participants affected / at risk) | 15/132 | 34/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=132) | Bimekizumab 160mg (N=267)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=132) | Bimekizumab 160mg (N=267)
Corona virus infection (Infections and infestations) | 6 (6) | 5 (5)
Nasopharyngitis (Infections and infestations) | 1 (1) | 10 (11)
Oral candidiasis (Infections and infestations) | 0 (0) | 7 (9)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 6 (6)
Urinary tract infection (Infections and infestations) | 3 (3) | 5 (6)
Hypertension (Vascular disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT03896581/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT03896581/SAP_001.pdf